CLINICAL TRIAL: NCT04206059
Title: Closed Loop Acoustic Stimulation During Sedation With Dexmedetomidine
Acronym: CLASS-D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ben J.A. Palanca, Assistant Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201907086
Record Dates: First submitted 2019-12-09; First posted 2019-12-20 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Sleep; Sedation Complication
MeSH Terms: interventions — Acoustic Stimulation; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CLASS-D Cohort (Experimental): Within-subject crossover cohort with intervention, acoustic stimulation delivered in phase with the anticipated trough of EEG slow wave oscillation, and 0 dB stimulation.
  Interventions: Radiation: MRI; Diagnostic Test: Quantitative Sensory Testing (QST); Diagnostic Test: Home sleep study; Other: Acoustic stimulation (65db) up-slope of EEG with QST; Other: Acoustic stimulation (65db) down-slope of EEG with QST; Other: 0 db with QST; Drug: Dexmedetomidine; Other: Breathe-Squeeze Task

INTERVENTIONS:
Radiation: MRI — A non-contrast brain MRI will be acquired for localizing EEG slow waves
  Other Names: Structural magnetic resonance imaging
Diagnostic Test: Quantitative Sensory Testing (QST) — Quantitative sensory testing (QST) using increasing ramp thermal stimulation (32-52 ºC) will be delivered to compare arousal thresholds between conditions.
  Other Names: Quantitative Sensory Testing
Diagnostic Test: Home sleep study — Unattended home sleep studies will be conducted on the night preceding sedation and on the night following sedation to assess changes in slow wave homeostasis.
  Other Names: Unattended polysomnography
Other: Acoustic stimulation (65db) up-slope of EEG with QST — Acoustic stimulation (65 db) synchronized in-phase with the up-slope of EEG slow waves
  Other Names: In-phase CLAS with sensory testing
Other: Acoustic stimulation (65db) down-slope of EEG with QST — 65 dB acoustic stimulation synchronized with the down-slope of the EEG slow waves (anti-phase)
  Other Names: Anti-phase CLAS with sensory testing
Other: 0 db with QST — sham stimulation (0 dB volume)
  Other Names: Sham CLAS with sensory testing
Drug: Dexmedetomidine — All participants will receive dexmedetomidine with sedation titrated step-wise to 2, 3 or 4 ng/ml
  Other Names: Dexmedetomidine hydrochloride
Other: Breathe-Squeeze Task — All participants will be asked to perform the breathe-squeeze task throughout the experiment. This will allow us to determine loss and return of responsiveness.
  Other Names: Internally directed behavioral task

SUMMARY:
Prospective within-subject study of dexmedetomidine sedation paired with CLAS conditions in repeated blocks. Intervention will consist of CLAS in-phase with EEG slow waves. Anti-phase stimulation will serve as an active control while sham stimulation will serve as a passive control.

DETAILED DESCRIPTION:
Both nonpharmacologic and pharmacologic interventions augment expression of EEG slow waves that mimic those of natural sleep. Closed loop auditory stimulation (CLAS) is a noninvasive inexpensive approach to augment the spectral power and duration of these slow waves. Whether in-phase CLAS may address this need is unknown, since acoustic potentiation of pharmacologically-induced slow waves has not been investigated. This prospective within-subject study of dexmedetomidine sedation paired with CLAS will assess the feasibility of augmenting EEG slow waves during sedation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Healthy volunteers (American Society of Anesthesiologists Physical Status 1-2).

Exclusion Criteria:

* Diagnosed sleep disorders
* Habitually short sleepers
* Diagnosed psychiatric disorders
* Use of psychoactive medication (e.g., antidepressants, mood stabilizers or antipsychotics), diagnosed hearing disorder
* Neck circumference > 40 cm
* Body Mass Index > 30
* Acknowledged recreational drug or nicotine use
* Resting heart rate during slow wave sleep < 40 beats per minute
* Pregnancy or nursing
* Persistently inconsistent or elevated QST heat pain tolerance thresholds (>50 ºC).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Difference in EEG slow wave amplitude from sham to in-phase stimulation | up to 3 months after consent
  EEG slow waves amplitude relative to the timing of the stimulation
Difference in EEG slow wave duration from sham to in-phase stimulation | up to 3 months after consent
  EEG slow waves duration relative to the timing of the stimulation
Difference in EEG slow wave amplitude from anti-phase to in-phase stimulation | up to 3 months after consent
  EEG slow waves amplitude relative to the timing of the stimulation
Difference in EEG slow wave duration from anti-phase to in-phase stimulation | up to 3 months after consent
  EEG slow waves duration relative to the timing of the stimulation

SECONDARY OUTCOMES:
Difference of reactivity to thermal stimulation from anti-phase to in-phase stimulation | up to 3 months after consent
  Threshold for responsiveness to thermal stimulation
Difference of reactivity to thermal stimulation from sham to in-phase stimulation | up to 3 months after consent
  Threshold for responsiveness to thermal stimulation
Change in slow wave activity on the night of the intervention will be compared to that on the night prior to the study session. | up to 3 months after consent
  Slow wave activity calculated during N3 sleep
Localization of slow waves | up to 3 months after consent
  Brain regions with localization of EEG slow waves during dexmedetomidine sedation

CONTACTS AND LOCATIONS:
Overall Officials: Ben J Palanca, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Prerau MJ, Brown RE, Bianchi MT, Ellenbogen JM, Purdon PL. Sleep Neurophysiological Dynamics Through the Lens of Multitaper Spectral Analysis. Physiology (Bethesda). 2017 Jan;32(1):60-92. doi: 10.1152/physiol.00062.2015. PMID 27927806
- [Background] Leger D, Debellemaniere E, Rabat A, Bayon V, Benchenane K, Chennaoui M. Slow-wave sleep: From the cell to the clinic. Sleep Med Rev. 2018 Oct;41:113-132. doi: 10.1016/j.smrv.2018.01.008. Epub 2018 Feb 5. PMID 29490885
- [Background] Neske GT. The Slow Oscillation in Cortical and Thalamic Networks: Mechanisms and Functions. Front Neural Circuits. 2016 Jan 14;9:88. doi: 10.3389/fncir.2015.00088. eCollection 2015. PMID 26834569
- [Derived] Smith SK, Kafashan M, Rios RL, Brown EN, Landsness EC, Guay CS, Palanca BJA. Daytime dexmedetomidine sedation with closed-loop acoustic stimulation alters slow wave sleep homeostasis in healthy adults. BJA Open. 2024 Mar 28;10:100276. doi: 10.1016/j.bjao.2024.100276. eCollection 2024 Jun. PMID 38571816
- [Derived] Guay CS, Hight D, Gupta G, Kafashan M, Luong AH, Avidan MS, Brown EN, Palanca BJA. Breathe-squeeze: pharmacodynamics of a stimulus-free behavioural paradigm to track conscious states during sedation☆. Br J Anaesth. 2023 May;130(5):557-566. doi: 10.1016/j.bja.2023.01.021. Epub 2023 Mar 24. PMID 36967282